CLINICAL TRIAL: NCT01554982
Title: A Long-Term Safety Extension Trial of KRX-0502 (Ferric Citrate) in Patients With End-Stage Renal Disease (ESRD) on Dialysis
Brief Title: A Long-Term Safety Extension Trial of Ferric Citrate in Patients With End-Stage Renal Disease (ESRD) on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRX-0502-307
Record Dates: First submitted 2012-03-12; First posted 2012-03-15 (Estimated); Results first posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-06

CONDITIONS: End Stage Renal Disease; Kidney Failure; Renal Failure; Hyperphosphatemia; ESRD
Keywords: Participation Limited; Long Term; Safety Extension
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Hyperphosphatemia | interventions — ferric citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ferric Citrate (Other): Open label extension of those completing study KRX-0304
  Interventions: Drug: ferric citrate

INTERVENTIONS:
Drug: ferric citrate — Dose based on monthly serum phosphorus levels with goal of 3.5-5.5 mg/dL for all patients.
  Other Names: Auryxia; KRX-0502

SUMMARY:
A long-term safety study of ferric citrate (KRX-0502) in renal failure patients who have completed study KRX-0502-304. Only patients who participated in the KRX-0502-304 trial may participate in this trial.

DETAILED DESCRIPTION:
This study was an open-label, 48-week safety extension of Study KRX-0502-304 (Study 304), to evaluate the safety of long-term use of KRX-0502 in subjects with ESRD for up to 2 years of cumulative exposure. Subjects who completed the Safety Assessment Period (SAP) and, if eligible, the Efficacy Assessment Period (EAP) of Study 304, independent of their assigned treatment arm in the SAP or EAP of Study 304, were eligible for participation in this long-term safety extension study. No new subjects were permitted to enter this study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-breast-feeding females who participated in the Safety Assessment Period (SAP), and if eligible, the Efficacy Assessment Period (EAP) of Study KRX-0502-304
2. Willing and able to give informed consent

Exclusion Criteria:

1. Subjects on KRX-0502 (ferric citrate) in KRX-0502-304 who were treatment failures in first period
2. Any subject in Study KRX-0502-304 SAP who early terminated from the trial
3. Any subject who participated in Study KRX-0502-304 but declined EAP
4. Actively symptomatic gastrointestinal bleeding or inflammatory bowel disease
5. History of malignancy in the last five years
6. Previous intolerance to KRX-0502 (ferric citrate)
7. Intolerance to oral iron-containing products
8. Absolute requirement for oral iron therapy
9. Absolute requirement for Vitamin C (multivitamins [Nephrocaps, Renaphro, etc.] allowed)
10. Absolute requirement for calcium-, magnesium-, or aluminum-containing drugs with meals
11. Inability to tolerate oral drug intake
12. Any other medical condition that rendered the subject unable to or unlikely to complete the trial or that would interfere with optimal participation in the trial or produce significant risk to the subject
13. Inability to cooperate with study personnel or history of noncompliance
14. Unsuitable for this trial per Principal Investigator's (PI) clinical judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia B Lewis, MD, Study Chair — Collaborative Study Group
Locations (34):
- United States (33):
  - Veterans Administration Greater Los Angeles Health Care System, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Western Nephrology and Metabolic Bone Disease, PC, Westminster, Colorado
  - Kidney Care Associates, LLC, Augusta, Georgia
  - Circle Medical Management, Chicago, Illinois
  - DaVita Dialysis Unit 494/Nephrology Specialists, PC, Michigan City, Indiana
  - Dept of Internal Medicine, Nephrology & Hypertension, New Orleans, Louisiana
  - Washington Nephrology Associates, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Western New England Renal & Transplant Associates, PC, Springfield, Massachusetts
  - Nephrology Hypertension Clinic, PC, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Rochester Hills DaVita Dialysis, Pontiac, Michigan
  - Asheville Kidney Center, Asheville, North Carolina
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - Duke University Dept of Medicine/Nephrology, Durham, North Carolina
  - Piedmont Dialysis Center, Winston-Salem, North Carolina
  - Clinical Research Limited, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Southeast Renal Research Institute Nephrology Associates, Chattanooga, Tennessee
  - Nephrology Associates, PC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Kidney Associates, PLLC, Houston, Texas
  - Med Center Dialysis, Houston, Texas
  - Kidney Specialists of North Houston, PLLC, Houston, Texas
  - University of Vermont/ Fletcher Allen Health Care: Renal Services, Burlington, Vermont
  - Nephrology Clinical Research Center, Charlottesville, Virginia
  - Clinical Research & Consulting Center, LLC, Fairfax, Virginia
  - Nephrology Associates of Northern Virginia, Inc., Fairfax, Virginia
  - Butler Farms Dialysis, Hampton, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- RCMI-Clinical Research Center, Rio Piedras, PR, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ferric Citrate
Started | 168
Received Drug | 166
Completed | 125
Not Completed | 43

BASELINE CHARACTERISTICS:
Population: Note: two subjects randomized did not receive study drug, therefore not included in Safety Assessment Population
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 135
  >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 103
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 2
  United States | 164

OUTCOME MEASURES:

1. Primary Outcome: Safety Parameters
Description: Safety was assessed by recording and monitoring adverse events (AEs), serious adverse events (SAEs), and sequential laboratory data. Rates of AEs were summarized by system organ class, preferred term, severity, and suspected relationship to KRX-0502 (ferric citrate).
Time Frame: 48 Weeks
Population: Safety Population; Treatment Emergent Adverse Events (TEAEs), not including SAEs, reported include only those occurring at a frequency >5%
Measure: Number; unit: participants
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 166
participants
  Subjects with at least 1 TEAE | 142
  Subjects with at least 1 related TEAE | 35
  Subjects with at least 1 serious TEAE | 75
  Subjects with at least 1 related, serious TEAEa | 0
  Total # of deaths | 10

2. Other Pre Specified Outcome: Serum Phosphorus- Baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 166
mg/dL | 5.7 (1.66)

3. Other Pre Specified Outcome: Serum Phosphorus- Week 48
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 126
mg/dL | 5.2 (1.34)

4. Other Pre Specified Outcome: Ferritin- Baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 166
ng/mL | 709.7 (385.11)

5. Other Pre Specified Outcome: Ferritin- Week 48
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 126
ng/mL | 821.0 (411.54)

6. Other Pre Specified Outcome: Transferrin Saturation (TSAT) - Baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 166
percentage of saturation | 32.4 (13.51)

7. Other Pre Specified Outcome: TSAT- Week 48
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 126
percentage of saturation | 40.3 (19.12)

8. Other Pre Specified Outcome: Hemoglobin- Baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 166
g/dL | 11.1 (1.36)

9. Other Pre Specified Outcome: Hemoglobin- Week 48
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 126
g/dL | 11.3 (1.38)

10. Other Pre Specified Outcome: IV Iron Use
Description: Percent of subjects with No IV iron intake from first dose of study drug to Week 48
Time Frame: 48 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Ferric Citrate
Number analyzed (Participants) | 166
percentage of participants | 59.0

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Treatment-emergent adverse events
Arm/Group | Ferric Citrate
Serious Adverse Events (participants affected / at risk) | 75/166
Other Adverse Events (participants affected / at risk) | 142/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Citrate (N=166)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (5)
Angina pectoris (Cardiac disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 6 (6)
Cardiac failure congestive (Cardiac disorders) | 4 (4)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleuropericarditis (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Dyspnoea (Cardiac disorders) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Death (General disorders) | 2 (2)
Necrosis (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 5 (5)
Sudden death (General disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Cellulitis streptococcal (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Incision site abscess (Infections and infestations) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (2)
Klebsiella bacteraemia (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Peritoneal abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 10 (10)
Postoperative wound infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 8 (8)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (2)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2)
Vascular graft complication (Injury, poisoning and procedural complications) | 2 (2)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (3)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Aspiration pleural cavity (Investigations) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Metabolic encephalopathy (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 4 (4)
Unresponsive to stimuli (Nervous system disorders) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1)
Catheter placement (Surgical and medical procedures) | 2 (2)
Leg amputation (Surgical and medical procedures) | 2 (2)
Parathyroidectomy (Surgical and medical procedures) | 1 (1)
Peritoneal dialysis (Surgical and medical procedures) | 1 (1)
Renal transplant (Surgical and medical procedures) | 10 (10)
Spinal fusion surgery (Surgical and medical procedures) | 1 (2)
Aneurysm (Vascular disorders) | 1 (1)
Brachiocephalic vein stenosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 2 (2)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 5 (6)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Abdominal Abscess (Infections and infestations) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Citrate (N=166)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 12 (17)
Constipation (Gastrointestinal disorders) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 26 (29)
Dizziness (Nervous system disorders) | 9 (13)
Dyspnoea (Cardiac disorders) | 13 (16)
Faeces discoloured (Gastrointestinal disorders) | 14 (14)
Fall (Injury, poisoning and procedural complications) | 9 (14)
Headache (Nervous system disorders) | 14 (23)
Hypertension (Vascular disorders) | 9 (11)
Hypotension (Vascular disorders) | 10 (66)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (16)
Nasopharyngitis (Infections and infestations) | 10 (11)
Nausea (Gastrointestinal disorders) | 17 (20)
Oedema peripheral (Gastrointestinal disorders) | 10 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (28)
Pyrexia (General disorders) | 9 (9)
Vascular graft complication (Injury, poisoning and procedural complications) | 9 (10)
Vomiting (Gastrointestinal disorders) | 16 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No